CLINICAL TRIAL: NCT05704491
Title: Accuracy of an AI Model for Diabetic Retinopathy Screening in Real-life
Brief Title: AI Screening for Diabetic Retinopathy
Acronym: AimdR
Status: Recruiting | Type: Observational
Sponsor: West German Center of Diabetes and Health (Other)
Responsible Party: Sponsor
Other Study IDs: AimdR
Record Dates: First submitted 2023-01-19; First posted 2023-01-30 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Artificial Intelligence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- K+A+: diabetic retinopathy according to AI present (K+) AND diabetic retinopathy according to the doctor present (A+)
  Interventions: Diagnostic Test: artificial intelligence (AI) algorithm of the MONA DR model
- K+A-: diabetic retinopathy according to AI present (K+) AND diabetic retinopathy according to the doctor absent (A-)
  Interventions: Diagnostic Test: artificial intelligence (AI) algorithm of the MONA DR model
- K-A+: diabetic retinopathy according to AI absent (K-) AND diabetic retinopathy according to the doctor present (A+)
  Interventions: Diagnostic Test: artificial intelligence (AI) algorithm of the MONA DR model
- K-A-: diabetic retinopathy according to AI absent (K-) AND diabetic retinopathy according to the doctor absent (A-)
  Interventions: Diagnostic Test: artificial intelligence (AI) algorithm of the MONA DR model

INTERVENTIONS:
Diagnostic Test: artificial intelligence (AI) algorithm of the MONA DR model — A 45-degree fundus image is taken for each eye and patient using the Crystalvue NFC 600. The fundus photographs are then analyzed using the MONA DR model and classified for presence of diabetic retinopathy.

SUMMARY:
The increasing prevalence of diabetes mellitus represents a major health problem, especially since around 40% of diabetic patients develop diabetic retinopathy, which severely impairs vision and can lead to blindness. This development could be prevented by annual check-ups and timely referral for treatment. However, there are major differences in the quality of examinations and bottlenecks in examination appointments. A solution to the problem could be the use of artificial intelligence (AI), especially deep learning. Initial studies have shown that deep learning algorithms can be used successfully to detect diabetic retinopathy. However, it remains to be clarified whether the use of AI can achieve a sufficiently high level of accuracy in the detection of retinopathies. Therefore, in the present study, the positive predictive value (PPV), the negative predictive value (NPV), the sensitivity (SEN) and the specificity (SPEZ) of the AI algorithm 'MONA-DR-Model' in the detection of diabetic retinopathy should be measured. In addition, it is to be examined how well the classification into mild and severe retinopathy corresponds and how well this new examination method is accepted by the patients.

DETAILED DESCRIPTION:
As part of the study, a 45-degree fundus image is taken for each eye and patient using the 'Crystalvue NFC 600'. The fundus photographs are then analyzed using the 'MONA-DR-Mode'l and classified as "diabetic retinopathy according to AI present (K+)" or "diabetic retinopathy according to AI absent (K-)". These classifications are compared with the results ("diabetic retinopathy according to the doctor present (A+)" or "diabetic retinopathy according to the doctor absent (A-)") of the examinations routinely provided for in the Disease Management Program (DMP) diabetes mellitus type 2 by resident ophthalmologists who work in the period 6 months before and after the fundus photography in the West German Centre of Diabetes and Health (WDGZ) were compared. All patients with the assessment "diabetic retinopathy according to AI present (K+)" or discrepancies with the ophthalmological DMP examination in the outpatient environment are offered a routine appointment at the Marienhospital. There, an eye examination is then carried out by an ophthalmologist and, without knowledge of the previous findings, a reassessment and classification as "diabetic retinopathy according to the doctor present (A+)" or "diabetic retinopathy according to the doctor absent (A-)" is carried out by the AI.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diabetes mellitus
* Diabetes duration ≥ 5 years
* Age > 18 years old
* Patient is able to give informed consent
* Fluent in written and spoken German, or interpreter present

Exclusion Criteria:

* History of laser treatment
* Contraindication to the fundus imaging systems used in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of the West German Centre of Diabetes and Health with Type 2 Diabetes
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-01-30 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
PPV | 12 months
  positive predictive value
NPV | 12 months
  negative predictive value
SEN | 12 months
  sensitivity
SPEZ | 12 months
  specificity

CONTACTS AND LOCATIONS:
Locations (1):
- West German Center of Diabetes and Health, Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: No